CLINICAL TRIAL: NCT05569265
Title: Open-label, Multicenter, Randomized, Controlled Trial of Hemodynamic Optimization Based on the Hypotension Prediction Index (HPI) Compared to Standard Practice in Adult Patients Undergoing Elective Major Abdominal Surgery.
Brief Title: Hypotension Prediction Index-guided Hemodynamic Optimization Trial to Reduce Postoperative Acute Kidney Injury (HYT).
Acronym: HYT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maria José Clara Colomina Soler (Other)
Responsible Party: Sponsor-Investigator, Maria José Clara Colomina Soler, Dr., Sociedad Española de Anestesiología, Reanimación y Terapéutica del Dolor
Organization: Sociedad Española de Anestesiología, Reanimación y Terapéutica del Dolor (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: GFMH1
Record Dates: First submitted 2022-10-04; First posted 2022-10-06 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Postoperative Acute Kidney Injury; Postoperative Complications
Keywords: Perioperative care; Acute kidney injury; Hemodynamic prediction index; Major surgery
MeSH Terms: conditions — Postoperative Complications; Acute Kidney Injury | interventions — Fluid Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hemodynamic prediction index based goal directed hemodynamic therapy (Experimental): Hemodynamic handling will be based hemodynamic prediction index (HPI)
  Interventions: Procedure: Intraoperative hemodynamic management
- No HPI (No Intervention): Patients in the control group will be treated according to standard practice.

INTERVENTIONS:
Procedure: Intraoperative hemodynamic management — Goal directed Hemodynamic therapy
  Other Names: Fluid therapy
  Arms: Hemodynamic prediction index based goal directed hemodynamic therapy

SUMMARY:
MAIN AIM OF THE STUDY To establish whether hemodynamic management guided by the hypotension prediction index (HPI) guided by the administration of intravenous fluids and vasoactive drugs in patients undergoing elective major abdominal surgery reduces the incidence of postoperative moderate-severe acute kidney injury (AKI) in the 30 days after surgery.

STUDY DESIGN A low intervention level clinical, blinded, controlled, randomized, multicenter, with daily follow-up of patients until hospital discharge and of postoperative complications and mortality 30 days after surgery will be performed.

This is a low-intervention clinical trial comparing standard treatments:

* The drugs used in the investigation are licensed.
* The drugs are used according to the indications contemplated in the technical data sheet and there are published scientific data on their efficacy and safety.
* The complementary diagnostic or follow-up procedures entail a very limited additional risk or burden to the safety of the subjects, which is minimal compared to that of standard clinical practice.

STUDY DISEASE Intraoperative hemodynamic monitoring and management in surgical patients undergoing major abdominal surgery.

STUDY POPULATION AND TOTAL NUMBER OF PATIENTS The sample of this study consists of patients of both genders, aged over 65 years and/or physical status ASA III or IV, undergoing elective major abdominal surgery (abdominal, urological, gynecological) under general/combined anesthesia (using laparoscopic or open approaches.

To detect a 5% absolute reduction (from 10% to 5%) in the primary outcome variable (postoperative AKI up to 30 days) with a sample size ratio of 1%, and an overall type I error rate of 5%, we need 870 patients (435 per arm). Assuming a 10% loss rate, the total amounts to 958 patients, 479 for each group.

DURATION OF THE STUDY The total planned duration of the overall study, which includes authorization, recruitment of subjects, and follow-up of subjects until completion of the analysis of the results obtained, is 19 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 65 years of age and/or physical condition ASA III or IV.
* Patients who have major elective abdominal surgery indicated: general surgery, urology, gynecology, by laparoscopic or open approaches.
* Patients who sign the informed consent, agreeing to participate in the study.

Exclusion Criteria:

* Stage 4 or 5 chronic kidney disease (eGFR < 15 ml/ min)
* Renal transplantation in the previous 12 months
* Glomerulonephritis, interstitial nephritis or vasculitis
* Anuria at inclusion
* Pre-existing AKI
* Renal replacement therapy (RRT) in the last 90 days
* Indication for renal replacement at the time of inclusion
* Participation in another interventional trial investigating a drug/intervention affecting renal function
* Patients with atrial fibrillation
* Patients with known cardiac shunts.
* Patients whose surgical indication is urgent
* Pregnancy or lactation
* Patients expected to die within 30 days.
* Acute myocardial ischemia within the previous 30 days.
* Acute pulmonary edema within the previous 30 days
* Any contraindication to vasoactive or inotropic medication at low doses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 958 (Actual)
Dates: Start 2022-10-08 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-02-25 (Actual)

PRIMARY OUTCOMES:
Acute kidney injury | 7 days after surgery
  The primary outcome is the occurrence of moderate or severe AKI (according to KDIGO Stage 2-3 criteria) within 30 days after surgery. AKI is classified according to the Kidney Disease: Improving Global Outcomes (KDIGO) criteria as follows:
  Stage 1: Increase in serum creatinine by 1.5 to 1.9 times baseline or increase in serum creatinine by 0.3 mg/dL, or reduction in urine output to <0.5 mL/kg/hour for 6 to 12 hours.
  Stage 2: Increase in serum creatinine by 2.0 to 2.9 times baseline, or reduction in urine output to <0.5 mL/kg/hour for >12 hours.
  Stage 3: Increase in serum creatinine to 3.0 times baseline, or increase in serum creatinine to >4.0 mg/dL or reduction in urine output to <0.3 mL/kg/hour for >24 hours, or anuria for >12 hours, or initiation of renal replacement therapy, or, in patients <18 years, decrease in estimated glomerular filtration rate (eGFR) to <35 mL/min/1.73 m2.

SECONDARY OUTCOMES:
Need for renal replacement therapy (RRT) | 30 days after surgery
  yes/no
renal replacement therapy (RRT) duration | 30 days after surgery
  days
Renal recovery on day 30 | 30 days after surgery
  yes/no
Mortality | 30 days after surgery
  yes/no
Postoperative complications | 30 days after surgery
  According to:Standards for definitions and use of outcome measures for clinical effectiveness research in perioperative medicine: European Perioperative Clinical Outcome (EPCO) definitions: a statement from the ESA-ESICM joint taskforce on perioperative outcome measures
Postoperative length of stay | 30 days after surgery
  days
Number of days free from critical care | 30 days after surgery
  days

CONTACTS AND LOCATIONS:
Overall Officials: Javier Ripollés Melchor, MD, Study Chair — Sociedad Española de Anestesiología, Reanimación y Terapéutica del Dolor
Locations (26):
- Spain (26):
  - Hospital Universitario Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario de Badajoz, Badajoz
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Universitario de Sant Pau, Barcelona
  - Hospital Universitario Moises Brogi, Barcelona
  - Hospital Uniuversitario de Basurto, Bilbao
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Universitario Doctor Trueta, Girona
  - Hospital San Cecilio, Granada
  - Hospital Universitario Virgen de Las Nieves, Granada
  - Hospital Universitario Juan Ramón Jimenez, Huelva
  - Hospital Universitario de Igualada, Igualada
  - Hospital Universitario Jerez de la Frontera, Jerez de la Frontera
  - Hospital Universitario de Gran Canaria Doctor Negrín, Las Palmas de Gran Canaria
  - Hospital Infanta Leonor, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario Puerta de Hierro, Majadahonda
  - Althai Xarxa Universitaria, Manresa
  - Hospital Universitario de Donostia, San Sebastián
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Clínico Universitario de Santiago, Santiago de Compostela
  - Hospital Universitario Virgen de la Macaarena, Seville
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital General Universitario de Valencia, Valencia
  - Hospital Universitario Ríio Hortega, Valladolid

IPD SHARING:
Plan to Share IPD: Yes
Upon specific request following the publication of the study
Supporting Information: Study Protocol, SAP, ICF
Time Frame: From publication on clinicaltrials.org until 1 year after publication of the results.
Access Criteria: under request and Steering Committe review

REFERENCES:
- [Background] Walsh M, Devereaux PJ, Garg AX, Kurz A, Turan A, Rodseth RN, Cywinski J, Thabane L, Sessler DI. Relationship between intraoperative mean arterial pressure and clinical outcomes after noncardiac surgery: toward an empirical definition of hypotension. Anesthesiology. 2013 Sep;119(3):507-15. doi: 10.1097/ALN.0b013e3182a10e26. PMID 23835589
- [Background] Wijnberge M, Geerts BF, Hol L, Lemmers N, Mulder MP, Berge P, Schenk J, Terwindt LE, Hollmann MW, Vlaar AP, Veelo DP. Effect of a Machine Learning-Derived Early Warning System for Intraoperative Hypotension vs Standard Care on Depth and Duration of Intraoperative Hypotension During Elective Noncardiac Surgery: The HYPE Randomized Clinical Trial. JAMA. 2020 Mar 17;323(11):1052-1060. doi: 10.1001/jama.2020.0592. PMID 32065827
- [Derived] Ripolles-Melchor J, Carrasco-Sanchez L, Tome-Roca JL, Aldecoa C, Zorrilla-Vaca A, Lorente-Olazabal JV, Colomina MJ, Perez A, Jimenez-Lopez JI, Navarro-Perez R, Abad-Gurumeta A, Monge-Garcia MI; HYT Study Group. Hypotension prediction index guided goal-directed therapy to reduce postoperative acute kidney injury during major abdominal surgery: study protocol for a multicenter randomized controlled clinical trial. Trials. 2024 Apr 29;25(1):288. doi: 10.1186/s13063-024-08113-w. PMID 38685032